CLINICAL TRIAL: NCT04987424
Title: Prevalence Of Upper Limb Lymphedema In Patients Diagnosed With Breast Cancer In A Valle Del Cauca Oncology Institution In A 2008-2020 Cohort In Colombia.
Brief Title: Prevalence of Lymphedema in Valle Del Cauca, Colombia.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grupo de investigación C.E.R (Other)
Collaborators: Hematooncologos S.A. (Unknown)
Responsible Party: Principal Investigator, Maria Isabel Cadena, Cirujana Plástica Estética, Reconstructiva y Microcirugía, Grupo de investigación C.E.R
Other Study IDs: CER2021
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Unilateral Breast Cancer
Keywords: Lymphedema; breast cancer; prevalence; risk factors; epidemiology
MeSH Terms: conditions — Unilateral Breast Neoplasms; Lymphedema; Breast Neoplasms | interventions — Growth and Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Development and validation of Lymphedema levels diagnostic — A single intervention was carried out in which the patients were summoned for an interview and anthropometric measurements of the upper limbs, thus calculating the arm volume for a lymphedema primary diagnosis .

SUMMARY:
This is an epidemiological cross-sectional study aiming to determine the prevalence of lymphedema and the incidence of risk factors in patients diagnosed with unilateral breast cancer in a cohort from 2008 to 2020 in a specialised oncology centre in Valle del Cauca, Colombia.

DETAILED DESCRIPTION:
CONTEXT: Breast cancer-associated lymphedema is considered one of the most frequent side effects of breast cancer therapy. (1,2) Despite the abundant information available worldwide on epidemiology and risk factors, little is known about these data in Colombia and Latin America.

OBJECTIVE: To determine the actual prevalence and incidence of risk factors for the development of lymphedema associated with breast cancer in a specialised oncology centre in Valle del Cauca, Colombia.

DESIGN, SETTING, AND PATIENTS: Between 2008 and 2020 a sample of 367 patients with a diagnosis of unilateral breast cancer was established, with which a descriptive study was carried out, in which a series of anthropometric measurements were taken of the upper limbs in order to obtain the volume of both arms and determine the prevalence of lymphedema using the formula of truncated volumes of the Spanish society of lymphology, after which the medical records were reviewed in order to collect other data of interest. Patients were excluded if they had bilateral breast cancer or direct trauma to the upper limb.

INTERVENTIONS: A single intervention was carried out in which the patients were summoned for an interview and anthropometric measurements of the upper limbs, thus calculating the arm volume for a lymphedema primary diagnosis .

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer, cancer diagnosis between 2008-2020 in the oncology institution Colombia

Exclusion Criteria:

* Moving to a different institution for attention (other than Hemato-Oncólogos SA), unwillingness to become volunteer and death, bilateral breast cancer, congenital disease or trauma in the upper limb.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 2008 and 2020 a sample of 367 patients with a diagnosis of unilateral breast cancer was established
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of lymphedema | 2014-2020
  Determining the prevalence of lymphedema in patients diagnosed with unilateral breast cancer

SECONDARY OUTCOMES:
Risk Factors | 2014-2020
  Determining risk factors for the development of lymphedema in patients diagnosed with unilateral breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Hematoncologos S.A, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- See also: Hematooncologos web page — https://hematooncologos.com/